CLINICAL TRIAL: NCT07380321
Title: Perioperative Ultrasonographic Assessment Of Diaphragmatic Function İn Pediatric Obstructive Sleep Apnea
Brief Title: Diaphragm Ultrasound İn Children With OSAS
Status: Recruiting | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Demet Altun, Professor, Istanbul University
Other Study IDs: 2024/2005
Record Dates: First submitted 2026-01-17; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea of Child
Keywords: Pediatric Sleep Questionnaire; diaphragm ultrasound; adenotonsillectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obstructive Sleep Apnea Group: Children with obstructive sleep apnea syndrome, defined by at least 8 "yes" responses out of 22 items on the Pediatric Sleep Questionnaire (PSQ), scheduled for adenotonsillectomy under general anesthesia.
- Control Group: Children without obstructive sleep apnea, defined by fewer than 8 "yes" responses out of 22 items on the Pediatric Sleep Questionnaire (PSQ), scheduled for elective non-airway-related otolaryngologic surgeries under general anesthesia.

SUMMARY:
This is a prospective observational study evaluating perioperative diaphragmatic function by ultrasonography in children aged 1-12 years undergoing elective surgery under general anesthesia.

Participants will be classified preoperatively based on the parent-completed Pediatric Sleep Questionnaire (PSQ). Children with suspected obstructive sleep apnea syndrome who are scheduled for adenotonsillectomy will form the study group, while children without clinical findings suggestive of obstructive sleep apnea who are scheduled for elective non-airway-related otolaryngologic surgeries will serve as controls.

Diaphragm ultrasound assessments will be performed before and after surgery in the supine position during spontaneous breathing. Measurements will include diaphragmatic thickness at end-inspiration and end-expiration, diaphragmatic thickening fraction, and diaphragmatic excursion during quiet and deep breathing.

The primary objective is to compare diaphragmatic excursion and thickening fraction between groups. Secondary objectives include evaluating the association between perioperative respiratory parameters, postoperative recovery, and diaphragm ultrasound measures.

DETAILED DESCRIPTION:
This prospective observational study is designed to evaluate perioperative diaphragmatic function using ultrasonography in pediatric patients undergoing elective surgery under general anesthesia. The study will be conducted in children aged 1-12 years who are followed at the Department of Otolaryngology of Istanbul University Istanbul Faculty of Medicine and are scheduled for surgery based on clinical indications.

A total of 60 children will be enrolled in the study in accordance with predefined inclusion and exclusion criteria. Participants will be classified into two groups based on the results of the parent-completed Pediatric Sleep Questionnaire (PSQ) administered preoperatively. A PSQ total score of ≥0.33 (at least 8 "yes" responses out of 22 items) will be considered indicative of suspected obstructive sleep apnea, and children scheduled for adenotonsillectomy will form the study group. Children with a PSQ total score of <0.33 and no clinical findings suggestive of obstructive sleep apnea who are scheduled for elective non-airway-related otolaryngologic surgeries will be included in the control group.

All patients will receive standardized perioperative anesthesia and surgical care. Diaphragmatic ultrasonographic assessments will be performed in the supine position during spontaneous breathing preoperatively and postoperatively. Diaphragmatic thickness will be assessed using a 4-15 MHz linear transducer placed perpendicular to the chest wall at the 7th-9th intercostal space along the right anterior axillary line; thickness will be measured at end-inspiration and end-expiration, and the diaphragmatic thickening fraction will be calculated. Diaphragmatic excursion will be evaluated using a 1-6 MHz convex transducer positioned in the right anterior subcostal region between the midclavicular and anterior axillary lines, and craniocaudal excursion will be recorded during quiet and deep breathing.

The primary objective of this study is to evaluate diaphragmatic function by comparing diaphragmatic thickening fraction between children with suspected obstructive sleep apnea and a control group. Secondary objectives include the assessment of diaphragmatic excursion, the evaluation of associations between diaphragmatic ultrasonography parameters and perioperative respiratory variables, and the assessment of postoperative recovery characteristics. In this context, the study aims to investigate the role of diaphragmatic ultrasonography as a noninvasive perioperative assessment tool for the evaluation of respiratory function and perioperative respiratory findings in children with suspected obstructive sleep apnea undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* Children aged 1 to 12 years
* Scheduled to undergo elective surgery under general anesthesia
* Written informed consent obtained from parents or legal guardians
* Availability of a completed pediatric sleep questionnaire (PSQ)

Exclusion Criteria:

* Patients younger than 1 year or older than 12 years
* Presence of a neuromuscular disease
* Use of medications that may affect neuromuscular function
* Diaphragmatic paralysis
* ASA physical status III-IV
* Refusal to participate in the study or failure to provide informed consent
* Body mass index (BMI) > 35 kg/m²

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 1-12 years who are followed at the Department of Otolaryngology of Istanbul University Istanbul Faculty of Medicine and are scheduled for surgery will be included in this study. Participants will be assessed preoperatively using the Pediatric Sleep Questionnaire (PSQ). Children who answer "yes" to at least 8 of the 22 items and are scheduled to undergo adenotonsillectomy will be assigned to the obstructive sleep apnea syndrome (OSAS) group, whereas children who answer "yes" to fewer than 8 items and are scheduled to undergo elective non-airway-related otolaryngologic surgery will be included in the control group. Only children with ASA physical status I-II who meet the inclusion and exclusion criteria and for whom informed consent has been obtained will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic Thickening Fraction (%) | Following premedication and prior to anesthesia induction, and within the first hour after surgery during the postoperative recovery period.
  Diaphragmatic thickening fraction will be calculated as (thickness at end-inspiration - thickness at end-expiration) / thickness at end-expiration × 100%, measured by ultrasound. The primary comparison will be between the OSAS group and the control group. Measurements will be assessed before and after surgery.

SECONDARY OUTCOMES:
Diaphragmatic Thickness at End-Inspiration (mm) | Following premedication and prior to anesthesia induction, and within the first hour after surgery during the postoperative recovery period.
  Diaphragmatic thickness at end-inspiration will be measured by ultrasonography. Values will be compared between the OSAS group and the control group, as well as between preoperative and postoperative measurements.
Perioperative Respiratory and Recovery Parameters | During surgery and for the duration of postoperative recovery.
  Perioperative respiratory and recovery parameters will be recorded, including oxygen saturation (SpO₂), end-tidal carbon dioxide (EtCO₂) values, Aldrete scores at recovery room admission and discharge, and length of stay in the recovery room. These parameters will be evaluated for associations with diaphragmatic ultrasonography measures and study group (OSAS vs control).
Diaphragmatic Thickness at End-Expiration (mm) | Following premedication and prior to anesthesia induction, and within the first hour after surgery during the postoperative recovery period.
  Diaphragmatic thickness at end-expiration will be measured by ultrasonography. Values will be compared between the OSAS group and the control group, as well as between preoperative and postoperative measurements
Diaphragmatic Excursion During Quiet Breathing (mm) | Following premedication and prior to anesthesia induction, and within the first hour after surgery during the postoperative recovery period.
  Craniocaudal diaphragmatic excursion during quiet tidal breathing will be measured by M-mode ultrasonography. Values will be compared between the OSAS group and the control group, as well as between preoperative and postoperative measurements.
Diaphragmatic Excursion During Deep Breathing (mm) | Following premedication and prior to anesthesia induction, and within the first hour after surgery during the postoperative recovery period.
  Craniocaudal diaphragmatic excursion during deep breathing will be measured by M-mode ultrasonography. Values will be compared between the OSAS group and the control group, as well as between preoperative and postoperative measurements.
Diaphragmatic Excursion Ratio (Quiet Breathing / Deep Breathing) | Following premedication and prior to anesthesia induction, and within the first hour after surgery during the postoperative recovery period.
  The ratio of diaphragmatic excursion during quiet breathing to diaphragmatic excursion during deep breathing will be calculated. Values will be compared between the OSAS group and the control group, as well as between preoperative and postoperative measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Furkan Kelebek, Resident, Principal Investigator — Istanbul University; Demet Altun, Professor, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Department of Anesthesiology, Istanbul, Fatih, Turkey (Türkiye)